CLINICAL TRIAL: NCT05265039
Title: Exploring Mechanisms of Massed Cognitive Processing Therapy: A Randomized Controlled Trial
Brief Title: Exploring Mechanisms of Massed Cognitive Processing Therapy
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rush University Medical Center (Other)
Responsible Party: Principal Investigator, Philip Held, Assistant Professor of Psychiatry, Rush University Medical Center
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 21082701
Record Dates: First submitted 2022-01-26; First posted 2022-03-03 (Actual); Last update posted 2025-11-13 (Actual); Status verified 2025-11

CONDITIONS: PTSD
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Relaxation Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cognitive Processing Therapy (CPT) (Experimental)
  Interventions: Behavioral: Cognitive Processing Therapy
- Relaxation Training (RT) (Active Comparator)
  Interventions: Behavioral: Relaxation Training

INTERVENTIONS:
Behavioral: Cognitive Processing Therapy — An evidence-based treatment for posttraumatic stress disorder (PTSD)
  Arms: Cognitive Processing Therapy (CPT)
Behavioral: Relaxation Training — Guided relaxation
  Arms: Relaxation Training (RT)

SUMMARY:
The overall goal of this randomized controlled trial with partial crossover is to compare the effectiveness of 1-week virtual massed Cognitive Processing Therapy (CPT) to 5-day virtual relaxation training (RT) with regard to their ability to reduce posttraumatic stress disorder (PTSD) symptoms. Specifically, this study is designed to 1) examine changes in PTSD symptoms during and following the respective intervention, and 2) explore possible psychological treatment mechanisms, including cognitive control, inhibition, self-efficacy, and memory, and 3) examine possible moderators of treatment success (e.g. neuropsychological factors).

ELIGIBILITY:
Inclusion Criteria:

Are fluent in English

* Have experienced a Criterion A traumatic event during their lifetime
* Have a PTSD diagnosis verified via the Clinician Administered PTSD Scale for DSM
* Are interested in receiving evidence-based treatment (CPT) for PTSD and able to attend either 10 therapy sessions over the course of one week (5 days) or are interested and able to complete 5 relaxation training sessions over the course of one week (5 days)
* Are willing and able to complete self-report measures and clinician-rated assessments at multiple time points over the course of the study
* Reside in the state of Illinois during the course of treatment

Exclusion Criteria:

1. The traumatic event occurred in the past month
2. They are currently suicidal or homicidal (i.e., plan and intent)
3. They have unmanaged psychosis or mania
4. They have not been on a stable dose of psychotropic medication for at least one month by the time of the baseline assessment
5. They have completed an evidence-based cognitive behavioral PTSD treatment (e.g., Cognitive Processing Therapy or Prolonged Exposure) in the past 3 months or are currently receiving an evidence-based PTSD treatment
6. They have an intellectual disability or significant cognitive impairment that would prevent them from engaging in CPT
7. They have a serious or unstable medical illness or instability for which hospitalization may be likely within the next year
8. They have an active substance use disorder (within the past 3 months) that would require immediate medical observation if substance use was discontinued (i.e., potential lethality)
9. They are involved with current legal actions related to the traumatic event that is anticipated to be targeted during treatment
10. They have a visual or auditory impairment that would prevent them from fully participating in study activities
11. Subjects who, at the time of consent, appear to have extenuating life circumstances (e.g., unstable housing, no internet access, etc.) which, in the judgement of the Principal Investigator, could affect the ability to deliver the intervention with fidelity

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2022-04-26 (Actual); Primary Completion 2025-09-30 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Clinician-Administered PTSD Scale for DSM | Through study completion, an average of 8 months
  Clinician-Administered Assessment of PTSD
PTSD Checklist for DSM-5 Criteria | Through study completion, an average of 8 months
  Self Report Measure for PTSD

CONTACTS AND LOCATIONS:
Locations (1):
- Rush University Medical Denter, Chicago, Illinois, United States